CLINICAL TRIAL: NCT00877682
Title: Regional Cryoablation for Localized Adenocarcinoma of the Prostate
Brief Title: Prostate Conformal Cryotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Endocare, Inc. (Industry); Gen-Probe, Incorporated (Industry); FirmaMed (Unknown); Envisioneering Medical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0244; NCI-2011-01340 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Prostate Tumor; Adenocarcinoma of the Prostate; PCA; Regional Prostate Cryoablation; Cryotherapy; Cryoablation; Health Related Quality of Life; HRQOL
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cryosurgery; Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cryotherapy (Experimental): Under general anesthetic using ultrasonic guidance, freezing (cryoablation) portion of prostate.
  Interventions: Procedure: Cryoablation

INTERVENTIONS:
Procedure: Cryoablation — Under general anesthetic using ultrasonic guidance, freezing (cryoablation) portion of prostate.
  Other Names: Cryotherapy

SUMMARY:
The goal of this clinical research study is to learn if using cryotherapy to treat only the part of the prostate that contains cancer is an effective treatment for prostate cancer. The safety of this treatment will also be studied. Researchers also want to learn if treating only the part of the prostate with cancer causes less impact on your quality of life than other types of therapies.

DETAILED DESCRIPTION:
Cryotherapy (also called cryoablation) is an FDA approved treatment for prostate cancer. It involves placing multiple needles within the prostate and freezing the prostate, which will destroy both the cancerous and normal prostate tissue in a very controlled manner. It is possible to treat less than the whole prostate by only freezing the area of the prostate known to contain the cancer.

For this study, cryotherapy will be performed in a way similar to whole prostate cryotherapy, except the entire prostate will not be frozen. For this study, only that portion of the prostate with the most prostate cancer and the upper half of the opposite side of location of the cancer in the prostate will be treated. All areas of cancer may not be treated.

Cryotherapy:

Cryotherapy is performed under general anesthetic in the operating room. An ultrasound probe is inserted into the rectum to monitor the tissue freezing. A urethral warmer is inserted into the bladder through the penis to maintain the health of the urethra.

Quality-of-Life Questionnaires:

You will complete quality-of-life questionnaires before the prostate biopsy, and then at 3, 6, 12, 18, 24, 30, and 36 months after cryotherapy. The questionnaires will ask about your general health and your urinary, bowel, and sexual functions. The questionnaire should take about 15 minutes to complete each time.

Digital Rectal Exams and PCA3 Testing:

Before your cryotherapy and again before the biopsies at Months 6, 18 and 36 you will have a digital rectal exam (feeling the prostate through your anus) to check the status of the disease. You will also have digital rectal exams at Months 48 and 60 to check the status of the disease.

Urine will be collected after each digital rectal exam. This sample will be tested for PCA3, which has been associated with prostate cancer.

Prostate Biopsies:

You will have additional prostate biopsies at 6, 18, and 36 months after cryotherapy. About 12 biopsies samples will be collected each time from the same locations as during the screening biopsy. If you have rising PSA levels or your doctor thinks it is necessary, you and your doctor will discuss the need additional biopsies at Months 48 and 60.

This is an investigational study. Cryotherapy is FDA approved for the destruction of tissue, including prostate tissue. For the treatment of prostate cancer, it is commonly used to treat the entire prostate gland. This study is investigational because only a part of the prostate gland will be treated, instead of the entire gland. Partial organ treatment with cryotherapy is common for treatment of kidney, liver, and skin lesions.

Up to 100 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically identified adenocarcinoma of the prostate by minimum 6 core prostate biopsy.
2. Serum PSA </= 10 ng/mL before prostate biopsy
3. Less than 50% of samples from one side of the prostate positive for prostate cancer.
4. No greater than 50% of a single core total length occupied by prostate cancer.
5. No dominant Gleason 4 component. (e.g.; 4+X is not allowed, but X+4 is eligible)
6. No Gleason 5 component (primary, secondary or tertiary).
7. Subjects may have contralateral positive prostate biopsy in a single core within the eligibility biopsy so long as the involvement of this core is 2mm or less and no Gleason 4 or Gleason 5 pattern exists. This is considered to be Non-Dominant (Contralateral) Tumor Burden and is not exclusionary.
8. In the case that the confirmatory biopsy fails to sample the tumor again, patients will be allowed to continue into the therapeutic phase using the laterality information obtained during the eligibility biopsy.

Exclusion Criteria:

1. Medical History or Concurrent Disease which in the investigators mind places the patient at significant preoperative risk or for which the investigator does not feel this therapy is appropriate. Investigator believes subject is unwilling or unable to comply with study protocol requirements.
2. AUASI (American Urologic Association Symptom Index) score >/=20
3. Active urinary tract infection
4. Active treatment with anticoagulant/anti-platelet agent that cannot be safely stopped at the time of prostate biopsy and cryotherapy.
5. Medical or surgical castration initiated before or after the eligibility biopsy.
6. Patient is unable to provide informed consent.
7. Patients will undergo base line bone scan prior to cryoablation to evaluate for regions of abnormal uptake before therapeutic intervention. Metastatic disease by bone scintigraphy is exclusionary. Bone scans performed within 12 months prior to study entry will be used for study base line purposes and will not need to be repeated, unless clinically indicated.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-04-06 (Actual); Primary Completion 2018-01-14 (Actual); Study Completion 2018-01-14 (Actual)

PRIMARY OUTCOMES:
Patient Response | 6 months
  Result of biopsy at 6 months after therapy. A failure event is either a Failure of Patient Selection or a Failure of Treatment.

CONTACTS AND LOCATIONS:
Overall Officials: John F. Ward, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org